CLINICAL TRIAL: NCT00539331
Title: A Two-Part Study in Japanese Patients With Advanced or Metastatic NSCLC. Open-Label Phase I to Assess the Safety & Tolerability of AZD2171 in Combination With Pac/Carb, Then a Phase II, Randomised, Double-Blind Study to Assess the Efficacy of Pac/Carb Alone and in Combination With AZD2171 and Pac/Carb
Brief Title: Phase I/II Study of AZD2171 in Combination With Paclitaxel/Carboplatin in Japanese Non-Small Cell Lung Cancer Patients
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Jane Robertson, MSD, AstraZeneca
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D8480C00040
Record Dates: First submitted 2007-10-02; First posted 2007-10-04 (Estimated); Last update posted 2011-06-01 (Estimated); Status verified 2011-05

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Non-small Cell Lung Cancer; NSCLC; AZD2171; Paclitaxel/Carboplatin; Non-small Cell Lung Cancer (NSCLC)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — cediranib; Paclitaxel; Carboplatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Placebo Comparator): Paclitaxel/Carboplatin
  Interventions: Drug: Paclitaxel; Drug: Carboplatin
- 2 (Experimental): Paclitaxel/Carboplatin + AZD2171
  Interventions: Drug: AZD2171; Drug: Paclitaxel; Drug: Carboplatin

INTERVENTIONS:
Drug: AZD2171 — oral tablet
  Other Names: cediranib; RECENTIN™
  Arms: 2
Drug: Paclitaxel — intravenous infusion
  Other Names: Taxol®
Drug: Carboplatin — intravenous injection
  Other Names: CBDCA; Paraplatin®

SUMMARY:
The National Cancer Institute of Canada Clinical Trials Group (NCIC-CTG) has informed AstraZeneca that the BR24 Phase II/III study of cediranib at 30mg in first line non-small cell lung cancer (NSCLC) will not continue into Phase III following the planned end of Phase II efficacy and tolerability analysis by the study's Data Safety Monitoring Committee. Although evidence of clinical activity was seen, there appeared to be an imbalance in toxicity and therefore the study was considered not to have met the pre-defined criteria for automatic continuation into Phase III. As the design of Study 040 is similar to that of Study BR24, AstraZeneca has suspended recruitment into Study 040.

ELIGIBILITY:
Inclusion Criteria:

* Having histologically or cytologically confirmed NSCLC
* Patients with previously untreated advanced/metastatic (Stage IIIB/IV) or postsurgery recurrent NSCLC
* WHO performance status 0-1

Exclusion Criteria:

* Untreated unstable brain or meningeal metastases
* Patient with inappropriate laboratory tests values
* Patient with poorly controlled hypertension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2007-09; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
PART A : Safety and tolerability of AZD2171 in combination with pac/carbo in patients with non-small cell lung cancer | Assessed at each visit during Part A
PART B : Assess the efficacy of AZD2171 by assessment of progression free survival (PFS) | time to progression

SECONDARY OUTCOMES:
PART A : To examine the effect of AZD2171 on the PK of carboplatin and paclitaxel | Assessed at each visit during Part A
PART B : To determine the efficacy of AZD2171 by assessment of overall response rate, change in tumour size and overall survival | time to death

CONTACTS AND LOCATIONS:
Overall Officials: Jane Robertson, Study Director — AstraZeneca; Masahiro Fukuoka, MD, Principal Investigator — Sakai hospital Kinki University School of Medicine; Xiaojin Shin, MD, Study Chair — AstraZeneca
Locations (2):
- Japan (2):
  - Research Site, Osaka
  - Research Site, Tokyo